CLINICAL TRIAL: NCT01470794
Title: A Phase 1 Ascending Dose Trial of Safety and Tolerability of Toca 511, a Retroviral Replicating Vector, Administered to Subjects at the Time of Resection for Recurrent High Grade Glioma & Followed by Treatment With Toca FC, Extended-Release 5-FC
Brief Title: Study of a Retroviral Replicating Vector Combined With a Prodrug to Treat Patients Undergoing Surgery for a Recurrent Malignant Brain Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-11-01
Record Dates: First submitted 2011-11-04; First posted 2011-11-11 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma
Keywords: GBM; HGG; High grade glioma; Malignant glioma; Grade III glioma; Grad IV glioma; glioma; glioblastoma; Grade IV astrocytoma; brain cancer; recurrent glioblastoma; AA; AOD; anaplastic astrocytoma; Anaplastic oligodendroglioma; Anaplastic oligoastrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Brain Neoplasms | interventions — vocimagene amiretrorepvec; Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Toca 511 vector/Toca FC prodrug
  Interventions: Biological: Toca 511 vector; Drug: Toca FC

INTERVENTIONS:
Biological: Toca 511 vector — All patients will receive Toca 511, a retroviral replicating vector that expresses the cytosine deaminase (CD) gene. CD converts the antifungal 5-FC to the anti-cancer drug 5-FU in cells that have been infected by the Toca 511 vector. Beginning approximately 6 weeks after administration of Toca 511, patients will begin courses of oral Toca FC at pre-specified intervals, depending on cohort, during the approximately 30 week study.
  Other Names: Toca 511, RRV, retroviral replicating vector; 5-FC, flucytosine, 5-fluorocytosine, Toca FC
Drug: Toca FC
  Other Names: flucytosine, 5-FC, 5-FC XR, Toca FC

SUMMARY:
This is a multicenter study evaluating the safety and tolerability of increasing doses of Toca 511, a retroviral replicating vector, injected into the resection cavity of patients with Grade III or Grade IV Gliomas who have elected to undergo surgical removal of their tumor. Approximately 6 weeks after injection of Toca 511, patients will begin an oral courses of Toca FC, an antifungal agent. These one week courses of Toca FC will be repeated during the approximately 30 week study. Two separate cohorts of patients treated with Toca 511 and Toca FC will also be evaluated with either of the following standard treatments for glioma: lomustine or bevacizumab. After completion of this study, all patients will be eligible for enrollment and encouraged to enter a long-term continuation protocol that enables additional Toca FC treatment cycles to be given, as well as permits the collection of long-term safety and survival data.

ELIGIBILITY:
Inclusion Criteria (must all be answered "Yes"):

* Has the patient given written informed consent?
* Is the patient between 18 years old and 80 years old inclusive?
* Has the patient had histologically proven HGG with recurrence or progression following initial definitive therapy(s) such as surgery with or without adjuvant radiation therapy and/or chemotherapy (confirmed by diagnostic biopsy or contrast-enhanced MRI and evaluable by Macdonald criteria)? Note if first recurrence of GBM is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field.
* Does the patient have a single, HGG tumor recurrence/progression that is ≤ 5 cm in its greatest dimension?
* Based on the pre-operative evaluation, is the tumor recurrence/progression a candidate for ≥ 80% resection?
* Has the patient elected not to undergo treatment with the Gliadel® wafer?
* Does the patient have a Karnofsky performance status ≥ 70?
* Does the patient have an absolute neutrophil count (ANC) ≥ 1500/mm3?
* Does the patient have an absolute lymphocyte count ≥ 500/mm3?
* Does the patient have a platelet count ≥ 100,000/mm3?
* Does the patient have a Hgb ≥ 10 g/dL?
* Does the patient have a normal PT/PTT? (subnormal PT/PTT acceptable)
* Does the patient have an estimated glomerular filtration rate of at least 50 mL/min (inclusive) by the Cockcroft-Gault formula?
* Does the patient have an ALT < 3 times the upper limit of the laboratory reference range and total bilirubin < 1.5 mg/dL?
* If the patient is a female of childbearing potential, has she had a negative serum pregnancy test within the past 21 days?
* Is the patient willing to use condoms for contraception for 6 months after receiving Toca 511 or until there is no evidence of the virus in his/her blood, whichever is longer. If the patient is a fertile female, is she willing to use contraception for at least 12 months?
* Is the patient willing and able to abide by the protocol?

Exclusion Criteria (must all be answered "No"):

* Has the patient received cytotoxic chemotherapy within the past 3 weeks (6 weeks for nitrosoureas) of the planned surgery date?
* Does the patient have, or has the subject had, within the past 4 weeks any infection requiring antibiotic, antifungal or antiviral therapy?
* Has the patient had a surgical procedure in the last 28 days or a surgical wound that is not healed?
* Does the patient have any bleeding diathesis, or must the subject take any anticoagulants, or antiplatelet agents, including NSAIDs that cannot be stopped for surgery?
* Does the patient have a history of allergy or intolerance to flucytosine?
* Is the patient HIV positive?
* Does the patient have any gastrointestinal disease that would prevent him or her from being able to ingest or absorb flucytosine?
* Has the patient received any investigational treatment within the past 30 days?
* Is the patient breast feeding?
* Has the patient received Avastin® (bevacizumab) for this recurrence/progression, or within the past 5 weeks?
* Does the patient have a history of prior malignancy, excluding basal or squamous cell carcinoma of the skin, with an expected survival of less than five years?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | 2 months
  Excluding nausea, vomiting and fatigue, any Grade 3 or higher non-hematologic toxicity or any Grade 4 or higher hematologic toxicity, felt to be related to Toca 511 or the Toca 511/Toca FC combination.

SECONDARY OUTCOMES:
Overall Survival of Subjects | Overall survival, Overall survival at 6 months (OS6), 9 months (OS9), and 12 months (OS12)
Progression Free Survival (PFS) of Subjects | PFS of subjects at 6 months (PFS-6)

CONTACTS AND LOCATIONS:
Overall Officials: Asha Das, MD, Study Director — Tocagen Inc.; Timothy Cloughesy, MD, NO, Principal Investigator — University of California, Los Angeles
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - Henry Ford Hospital, Detroit, Michigan
  - JFK Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Swedish Neuroscience Institute, Seattle, Washington

REFERENCES:
- [Background] Ostertag D, Amundson KK, Lopez Espinoza F, Martin B, Buckley T, Galvao da Silva AP, Lin AH, Valenta DT, Perez OD, Ibanez CE, Chen CI, Pettersson PL, Burnett R, Daublebsky V, Hlavaty J, Gunzburg W, Kasahara N, Gruber HE, Jolly DJ, Robbins JM. Brain tumor eradication and prolonged survival from intratumoral conversion of 5-fluorocytosine to 5-fluorouracil using a nonlytic retroviral replicating vector. Neuro Oncol. 2012 Feb;14(2):145-59. doi: 10.1093/neuonc/nor199. Epub 2011 Nov 9. PMID 22070930
- [Derived] Cloughesy TF, Landolfi J, Vogelbaum MA, Ostertag D, Elder JB, Bloomfield S, Carter B, Chen CC, Kalkanis SN, Kesari S, Lai A, Lee IY, Liau LM, Mikkelsen T, Nghiemphu P, Piccioni D, Accomando W, Diago OR, Hogan DJ, Gammon D, Kasahara N, Kheoh T, Jolly DJ, Gruber HE, Das A, Walbert T. Durable complete responses in some recurrent high-grade glioma patients treated with Toca 511 + Toca FC. Neuro Oncol. 2018 Sep 3;20(10):1383-1392. doi: 10.1093/neuonc/noy075. PMID 29762717